CLINICAL TRIAL: NCT04195399
Title: A Safety, Pharmacokinetic and Efficacy Study of a y-Secretase Inhibitor, Nirogacestat (PF-03084014), in Children and Adolescents With Progressive, Surgically Unresectable Desmoid Tumors
Brief Title: A Study of a New Drug, Nirogacestat, for Treating Desmoid Tumors That Cannot be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARST1921; NCI-2019-07498 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST1921 (Other: Children's Oncology Group); ARST1921 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-12-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Desmoid Fibromatosis; Recurrent Desmoid Fibromatosis; Unresectable Desmoid Fibromatosis
MeSH Terms: conditions — Desmoid Tumors | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; nirogacestat; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (nirogacestat) (Experimental): Patients receive nirogacestat PO BID on days 1-28. Cycles repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO and CT or MRI on study. Patients may also undergo x-ray imaging and blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Drug: Nirogacestat; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Nirogacestat — Given PO
  Other Names: (S)-2-(((S)-6,8-Difluoro-1,2,3,4-tetrahydronaphthalen-2-yl)amino)-N-(1-(2-methyl-1-(neopentylamino)propan-2-yl)-1H-imidazol-4-yl)pentanamide; PF 03084014; PF-03084014; PF03084014
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial studies the side effects and how well nirogacestat works in treating patients less than 18 years of age with desmoid tumors that has grown after at least one form of treatment by mouth or in the vein that cannot be removed by surgery. Nirogacestat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 2-year progression-free survival (PFS) rate in patients with progressive, surgically unresectable desmoid tumor treated with nirogacestat.

II. To describe the toxicities of nirogacestat in children and adolescents with desmoid tumor.

III. To characterize the pharmacokinetics (PK) of nirogacestat in children and adolescents.

SECONDARY OBJECTIVE:

I. To determine the objective tumor response rate (ORR) of nirogacestat in children and adolescents with progressive, surgically unresectable desmoid tumor.

EXPLORATORY OBJECTIVES:

I. To collect blood, archival tumor samples and on-study/post-treatment tumor samples (if available) from patients enrolled on this trial to correlate various CTNNB1 and APC gene mutations and genomic signatures with tumor response and PFS.

II. To explore the effect of nirogacestat on immune cells and immunoglobulin levels in the peripheral blood.

III. To collect blood samples for banking at baseline, during treatment, and at the time of progression for future research.

IV. To compare assessment of tumor response using Response Evaluation Criteria in Solid Tumors (RECIST), World Health Organization (WHO) criteria, and T2 and volumetric changes using magnetic resonance imaging (MRI).

V. To utilize a tool developed to specifically assess patient reported outcomes (PROs) in adult patients with desmoid tumor (GOunder/DTRF DEsmoid Symptom/Impact Scale [GODDESS]) and the Patient Reported Outcomes Measurement Information System (PROMIS) to explore the relationship between PROs and tumor response and PFS.

OUTLINE:

Patients receive nirogacestat orally (PO) twice daily (BID) on days 1-28. Cycles repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) and computed tomography (CT) or MRI on study. Patients may also undergo x-ray imaging and blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 12 months and < 18 years of age at the time of enrollment
* Patients must have a body surface area of > 0.3 m^2 at the time of enrollment
* Existing or recurrent desmoid tumor that is deemed not amenable to surgery without significant morbidity and progressed by >= 10% as assessed by RECIST version (v)1.1 within the 6-month period prior to study enrollment

  * Patients must have had histologic verification of the desmoid tumor
  * Patients must have measurable disease by RECIST v1.1 criteria
  * Patient must have received at least one prior course of systemic therapy for desmoid tumor
* Patients must have a Lansky (for patients =< 16 years of age) or Karnofsky (for patients > 16 years of age) performance status score of >= 50. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, surgery or radiotherapy prior to entering this study. Patients may not be using or anticipate using these treatments after the observed progression or within the time period stated below

  * Cytotoxic chemotherapy: must not have received within 2 weeks of entry onto this study (4 weeks if prior nitrosourea)
  * Small molecule tyrosine kinase inhibitors (e.g., sorafenib, pazopanib, imatinib), rapalogs (e.g., temsirolimus, everolimus, sirolimus) or anti estrogen therapy (e.g., tamoxifen): may not have received within 28 days prior to the first dose of study treatment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent
  * Local regional tumor directed therapy, including, but not limited to small port radiation therapy (RT), radiofrequency ablation, cryotherapy, surgery: at least 2 weeks since these therapies and all toxicity must have resolved to grade =< 1. If prior craniospinal RT or if >= 50% radiation of pelvis then >= 6 months must have elapsed. If other substantial bone marrow (BM) radiation, then >= 6 weeks must have elapsed
  * Stem cell transplant (SCT): No evidence of active graft versus (vs.) host disease. For allogeneic SCT, >= 6 months must have elapsed
  * No prior gamma-secretase, Notch or beta-catenin inhibitor
  * Investigational drugs: must not have received investigational drug within 4 weeks of study entry, and all toxicities related to prior therapy must be resolved to grade =< 1 or baseline
* Concomitant Medication Restrictions

  * Growth factor(s): must not have received within 1 week of entry onto this study
  * Patients who are currently receiving drugs that are strong inducers or moderate or strong inhibitors of CYP3A4 are not eligible. Strong inducers or moderate or strong inhibitors of CYP3A4 are not allowed from 14 days prior to enrollment to the end of protocol therapy. Note: CYP3A4 inducing anti-epileptic drugs on a stable dose, are allowed
  * Must not be receiving non-steroidal anti-inflammatory drugs (NSAIDs) as treatment for desmoid tumor after the observed progression and patient agrees to not use NSAIDs while on study. Occasional use (defined as =< 3 times per week) for treatment of pain is permitted
* Peripheral absolute neutrophil count (ANC) >= 1000/uL (within 7 days prior to enrollment)
* Platelet count >= 100,000/uL (transfusion independent) (within 7 days prior to enrollment)
* Hemoglobin >= 9.0 g/dL (may receive red blood cell [RBC] transfusions) (within 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age: Maximum serum creatinine (mg/dL)
  * Age: 1 to < 2 years; Maximum serum creatinine (mg/dL): 0.6 (male and female)
  * Age: 2 to < 6 years; Maximum serum creatinine (mg/dL): 0.8 (male and female)
  * Age: 6 to < 10 years; Maximum serum creatinine (mg/dL): 1 (male and female)
  * Age: 10 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male and female)
  * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: >= 16 years; Maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)
* Adequate liver function defined as:
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (unless secondary to previously diagnosed Gilbert's syndrome) (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L (within 7 days prior to enrollment)
* Adequate cardiac function defined as:

  * Corrected QT (QTc) interval < 470 ms
  * No history of congenital or acquired prolonged QTc syndrome
  * No history of clinically significant cardiac arrhythmias, congestive heart failure, stroke or myocardial infarction within 6 months prior to study entry
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Active or chronic infection within 7 days prior to study entry
* Presence of non-healing fracture

  * Note: patients with pathologic fracture related to tumor are eligible
* Use of corticosteroids within 21 days of enrollment, except in the following situations:

  * Physiologic steroid replacement for adrenal insufficiency
  * Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
  * Short course (=< 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen), or exacerbation of asthma
* Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication, prior surgical procedures affecting absorption (e.g., gastric bypass), malabsorption syndrome, and active peptic ulcer disease)
* Patients with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction
* Known active infection with hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Patients with a prior history of malignancy, with the exceptions of desmoid tumor(s) and non-melanoma skin cancer, who are not in remission for more than 3 years
* Patients who are unable to swallow tablets. Tablets must not be crushed or chewed. Administration of nirogacestat via gastrostomy tube or nasogastric tube is not allowed
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study
* Sexually active female patients of reproductive potential who have not agreed to use 1 method of highly effective contraceptive (including copper-containing intrauterine device, condom with spermicidal foam/gel/film/cream/suppository, bilateral tubal ligation, established use of inserted, injected or implanted hormonal method of contraception, abstinence, or male sterilization) for the duration of their study participation and for at least 6 months after last dose of nirogacestat. A second form of contraception (i.e. barrier method) is required for patients who are using hormonal contraception as nirogacestat may reduce the efficacy of hormonal contraceptives
* Sexually active male patients of reproductive potential who have not agreed to use a condom and their female partner who have not agreed to use one of the highly effective methods of contraception mentioned above during treatment and for at least 90 days after the last dose of nirogacestat
* Female patients who are breastfeeding
* Female patients who are pregnant. These patients are excluded because there is no available information regarding the effects of nirogacestat on the developing human fetus and inhibition of gamma-secretase is known to be teratogenic
* Female patients of childbearing potential unless a negative pregnancy test result has been obtained

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From initiation of treatment to occurrence of disease progression or death from any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method with the 95% confidence interval estimated by the Peto-Peto method.
Incidence of adverse events | Up to 2 years
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All grade 3 or above toxicities deemed related to study drug will be summarized. All grade 1 and 2 toxicities observed in > 5% of participants and deemed related to study drug will be reported.
Pharmacokinetic (PK) parameter: systemic exposure | Up to Cycle 3 (each cycle lasts 28 days)
  PK parameters of nirogacestat will be defined to quantify systemic exposure, drug clearance, terminal half-life and other pharmacokinetic characteristics. These PK parameters will be summarized with descriptive statistics, including means, medians, ranges, and standard deviations.
PK parameter: drug clearance | Up to Cycle 3 (each cycle lasts 28 days)
  PK parameters of nirogacestat will be defined to quantify systemic exposure, drug clearance, terminal half-life and other pharmacokinetic characteristics. These PK parameters will be summarized with descriptive statistics, including means, medians, ranges, and standard deviations.
PK parameter: half-life | Up to Cycle 3 (each cycle lasts 28 days)
  PK parameters of nirogacestat will be defined to quantify systemic exposure, drug clearance, terminal half-life and other pharmacokinetic characteristics. These PK parameters will be summarized with descriptive statistics, including means, medians, ranges, and standard deviations.

SECONDARY OUTCOMES:
Objective response rate | Up to 24 months
  Defined by the rate of a complete response or partial response by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

OTHER OUTCOMES:
CTNNB1 and APC gene mutations and genomic signatures | Up to 2 years
  The chi-square test will be used to assess the correlation of CTNNB1 and APC gene mutations and genomic signatures with tumor response, and the long-rank test will be used to assess the correlation of CTNNB1 and APC gene mutations and genomic signatures with PFS.
Changes in the levels of each of the lymphocyte subsets and immunoglobulins | Up to 2 years
  Lymphocyte subsets include CD3 (total T cells), CD3+CD4+ (T helper cells), CD3+CD8+ (T cytotoxic cells), CD3+HLA-DR+ (activated T cells) percentages and absolute counts and CD4:CD8 ratio. The chi-square test will be used to assess the correlation of the levels of lymphocyte and immunoglobulin with tumor response, and the Cox regression will be used to assess the correlation of the levels of lymphocyte and immunoglobulin with PFS.
Response assessments by the RECIST criteria | Up to cycle 24
Response assessment by the World Health Organization criteria | Up to cycle 24
Patient reported outcomes (PROs) | Up to 2 years
  The chi-square test will be used to assess the correlation of PROs summary scores with tumor response, and the Cox regression will be used to assess the correlation of PROs summary scores with PFS. Correlation between PRO summary scores using Patient Reported Outcomes Measurement Information System and GOunder/DTRF DEsmoid Symptom/Impact Scale will be assessed by performing inferences on the Pearson correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Navid, Principal Investigator — Children's Oncology Group
Locations (98):
- United States (89):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Children's, Roanoke, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- University Pediatric Hospital, San Juan, Puerto Rico